CLINICAL TRIAL: NCT05744089
Title: A Single-arm Multicenter Study on the Home Management of Simple Hydromorphone PCA Pump Mode in Cancer Patients Suffering Severe or Critically Painful
Brief Title: Home Management of Simple Hydromorphone PCA Pump Mode
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCA001
Record Dates: First submitted 2023-02-13; First posted 2023-02-24 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Cancer Pain; Tumor, Solid; Carcinoma
MeSH Terms: conditions — Cancer Pain; Neoplasms; Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer patients suffering severe or critically painful (Experimental)
  Interventions: Device: PCA pump

INTERVENTIONS:
Device: PCA pump — simple hydromorphone PCA pump model, which is a rapid titration followed by a convenient maintenance technique, to treat home cancer patients with severe or critical cancer pain or refractory cancer pain.

SUMMARY:
This prospective observational study will evaluate the efficacy and adverse effects of a "simple hydromorphone PCA pump model", which is a rapid titration followed by a convenient maintenance technique, to treat home cancer patients with severe or critical cancer pain or refractory cancer pain.

DETAILED DESCRIPTION:
This is a single-arm multicenter study that will involve 8-10 centers and 50 cases in total. A better pumping mode was discovered through repeated optimization and adjustment of PCA pump parameters, ensuring the unity of convenience, safety, and flexibility: on the one hand, it is convenient for clinicians to set up and adjust the pump quickly; on the other hand, it is also convenient for patients to control at home; thus, it solves the complex pumping and dosing problems. Nearly 20 patients with severe cancer pain or a cancer pain crisis were treated using this model, and the control satisfaction rate was 100% in each case.

The purpose of this study is to:

1. Main objective: To explore the efficacy and adverse effects of a simple hydromorphone PCA pump model, i.e., rapid titration followed by maintenance, for the treatment of patients with severe cancer pain or cancer pain crisis or refractory cancer pain in home cancer patients.
2. Exploratory purpose: To screen sensitive indicators for cancer pain assessment and efficacy monitoring by Ella fully automated microfluidic ELISA system, and to explore the mechanism of action of pain-causing substances in cancer pain initially.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patients with pathologically confirmed malignant solid tumors; patients with advanced metastatic cancer assessed by imaging
3. Patients with persistent cancer pain and an NRS score of ≥7 in the past 24 hours; or patients with refractory pain
4. Patients who have not received radiation therapy within 7 days prior to randomization and trial
5. Patients without cognitive impairment or mental illness.
6. the patient is able to complete the survey form
7. Patients can correctly understand and cooperate with the healthcare provider's medication instructions.
8. ECOG-PS ≤ 3 points.
9. Subjects voluntarily and signed the informed consent form.
10. Failure of antineoplastic treatment or refusal of antineoplastic treatment at home or community hospital.

Exclusion Criteria:

1. Patients with a diagnosis of non-cancerous pain or pain of unknown origin.
2. Patients receiving inpatient antineoplastic therapy.
3. patients with paralytic intestinal obstruction
4. patients with opioid allergy.
5. abnormal and clinically significant laboratory results, such as creatinine ≥ 2 times the upper limit of normal, ALT or AST ≥ 2.5 times the upper limit of normal (≥ 5 times the upper limit of normal in patients with liver metastases or primary hepatocellular carcinoma), or grade C liver function Child
6. Uncontrollable nausea and vomiting.
7. Use of monoamine oxidase inhibitors within 14 days prior to randomization.
8. pregnant or lactating women; subjects with a planned pregnancy within 1 month of trial (also includes male subjects)
9. Patients with alcohol abuse.
10. Other diseases and conditions that, in the opinion of the investigator, preclude enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Pain score | 10 days
  Subjects self-assess on the NRS pain rating scale in the subject log sheet, where subjects assess the level of cancer pain experienced in the past 24 hours.
The frequency of paroxysmal pain | 10 days
  Paroxysmal pain is defined as a sudden and transient pain exacerbation that occurs spontaneously or triggered by some predictable or unpredictable factors under the premise of relatively stable background pain control and adequate application of analgesic drugs. The onset, duration and number of cancer eruption pain episodes were recorded by the subjects in the logbook at the time of the episode.
Life quality | 10 days
  The WHOQOL-BREF is a 26-item self-assessment questionnaire that investigates the last two weeks of physical health, mental health, social relationships, and environment. It allows for a reliable, valid and brief assessment of quality of life. In this study, the psychological domain (6 items) was used to represent the psychological aspects of quality of life.
The evaluation of PCA home feasibility | 10 days
  During the trial, monitoring the number of occurrences of PCA blockage and reflux in patients, as well as will record the number of times they seek help from healthcare professionals in case of PCA pump-related problems that cannot be solved by themselves.

SECONDARY OUTCOMES:
The concentration of immune-related cytokines | 10 days
  the content of PD 1, IL-2, IL-6, STING, CD3+, CD4+, IFN-1and IFN-γ in patients' serum

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided